CLINICAL TRIAL: NCT03449966
Title: Comparison of Ability of pCLE and WLE for Diagnosis and Cancer Tissue Acquisition in Advanced Gastric Cancer After Chemotherapy Status
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2017-0770
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Advanced Gastric Cancer; Neoadjuvant Chemotherapy; Palliative Chemotherapy
Keywords: pCLE; confocal; Advanced gastric cancer; chemotherapy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: All procedures were performed with both WLE and pCLE. One patient underwent both WLE and pCLE. Target biopsy under pCLE and random biopsy at cancer lesion under WLE will be done for one patient. The proportion of remnant cancer cells in biopsy samples will be compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Target biopsy under pCLE (Experimental): (Cellvisio® with confocal minoprobe™, Mauna Kea Technologies, France)
  Interventions: Device: Confocal group
- Random biopsy at cancer lesion under WLE (Active Comparator): WLE (GIF-HQ290, Olympus, Japan) group
  Interventions: Device: Control group

INTERVENTIONS:
Device: Confocal group — Under pCLE, target biopsy at cancer lesion will be done. 5 pieces of forcep biopsy will be obtained.
  Other Names: pCLE group
  Arms: Target biopsy under pCLE
Device: Control group — Random biopsy around cancer lesion will be done under WLE. 5 pieces with forcep biopsy will be obtained.
  Arms: Random biopsy at cancer lesion under WLE

SUMMARY:
* single center, prospective study First, evaluate the lesion under the white light endoscopy (WLE) → IV fluorescein sodium 0.1mL/kg → evaluate the lesion under probe-based confocal laser microendoscopy → target biopsy under the pCLE → random biopsy under WLE

DETAILED DESCRIPTION:
The purpose of this study is to conduct a study on genetic pathology, obtaining of cancer tissues is mandatory. Although the endoscopy with biopsy has been a gold standard for diagnosing gastric cancer, percentage of cancer cells in biopsy samples of patients after chemotherapy is usually 30% or less. Because cancer cells are often replaced with regenerative cells after chemotherapy, even though there are still remnant cancer cells in the stomach. Recently, confocal laser endomicroscopy has been introduced for real-time histopathologic diagnosis in various cancers. In previous pilot study in our institution, pCLE-targeted biopsy provided superior results in terms of the proportion of cancer cells in biopsy samples compared to WLE-targeted biopsy, especially for gastric cancers with undifferentiated histology. However, there was no previous study about precious biopsy method for patients after chemotherapy. Therefore, the investigators aim to evaluate that biopsy using probe-based confocal laser endomicroscopy for remnant gastric cancer after chemotherapy will increase the percentage of cancer cells and expression ratio of tumor marker in biopsy samples.

ELIGIBILITY:
Inclusion Criteria:

A. Older than 20 years old and younger than 80 years old B. Patients who completed neoadjuvant chemotherapy with AGC C. Patients who underwent palliative chemotherapy with AGC

Exclusion Criteria:

A. Previous subtotal gastrectomy B. Previous EMR/ESD history C. Significant cardiopulmonary disease D. Active hepatitis or severe hepatic dysfunction E. Severe renal dysfunction F. Severe bone marrow dysfunction G. Severe neurologic or psychotic disorder H. Pregnancy or breast feeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
The percentage of remnant cancer cells in biopsy samples | within the first day after pCLE
  The percentage of remnant cancer cells in biopsy samples according to the method of endoscopic method, probe-based confocal laser endomicroscopy versus white light endoscopy

SECONDARY OUTCOMES:
pCLE findings of residual cancer cells after chemotherapy | within the first day after pCLE
  The specific findins of remnant cancer cells under probe-based confocal laser endomicroscopy (ex. Destruction of gland structure, increased numbers of blood vessel, dark cells…)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university of medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No